CLINICAL TRIAL: NCT02474342
Title: Safety and Efficacy of Autologous Adipose Tissue Derived Mesenchymal Stem Cells Transplantation in Patient With Rotator Cuff Disease
Brief Title: Autologous Adipose Tissue Derived Mesenchymal Stem Cells for Rotator Cuff Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyunchul Jo, Associate Professor, SMG-SNU Boramae Medical Center, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRM-15-01
Record Dates: First submitted 2015-06-02; First posted 2015-06-17 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2016-05

CONDITIONS: Rotator Cuff Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous Adipose Tissue derived MSCs (Experimental)
  Interventions: Biological: Autologous Adipose Tissue Derived MSCs Transplantation

INTERVENTIONS:
Biological: Autologous Adipose Tissue Derived MSCs Transplantation — 1. Study drugs: Autologous adipose tissue derived MSCs
  2. Injection dosage and volume of the study drugs:
     * Low dose: 1x10e7 cells/3mL
  3. Number of injections : only once during the study period
  4. Device: Ultrasound
  5. Injection technique: Injection into the lesion by investigator
Biological: Autologous Adipose Tissue Derived MSCs Transplantation — 1. Study drugs: Autologous adipose tissue derived MSCs
  2. Injection dosage and volume of the study drugs:
     * Mid dose: 5x10e7 cells/3mL
  3. Number of injections : only once during the study period
  4. Device: Ultrasound
  5. Injection technique: Injection into the lesion by investigator
Biological: Autologous Adipose Tissue Derived MSCs Transplantation — 1. Study drugs: Autologous adipose tissue derived MSCs
  2. Injection dosage and volume of the study drugs:
     * High dose: 1x10e8 cells/3mL
  3. Number of injections : only once during the study period
  4. Device: Ultrasound
  5. Injection technique: Injection into the lesion by investigator

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of Autologous Adipose Tissue Derived Mesenchymal Stem Cells injection in patient with Rotator Cuff disease.

ELIGIBILITY:
Participants should meet all the inclusion criteria. Patients must consent in writing to participate in the study by signing and dating an informed consent document approved by IRB indicating that the patient has been informed of all pertinent aspects of the study prior to completing any of the screening procedures

Inclusion Criteria:

1. Male or female 19 years of age and older.
2. Patients who have unilateral shoulder pain.
3. Patients who have had pain at least for 3 months and do not respond to conservative treatment.
4. Patients who have a partial-thickness rotator cuff tear confirmed with magnetic resonance imaging (MRI) or ultrasonography (US).

Exclusion Criteria:

Participants who met a single condition were excluded from the study

1. Patients who received any drug by subacromial injection for treatment within 3 months prior to this enrollment.
2. Patients who have a history of shoulder trauma including dislocation, subluxation, and fracture, breast cancer, or surgery around shoulder, neck and upper back within 6 months prior to this enrollment.
3. Patients who have a full-thickness rotator cuff tear
4. Patients who have radiological findings of malignancy, osteoarthritis of the glenohumeral joint, and skeletal abnormalities decreasing the subacromial space
5. Patients with symptomatic cervical spine disorders
6. Patients with concurrent bilateral shoulder pain
7. Patients with adhesive capsulitis, acromioclavicular arthropathy, polyarthritis, infectious arthritis, rheumatoid arthritis or diagnosed fibromyalgia
8. Patients with neurological deficit
9. Pregnant women or lactating mothers
10. Fertile woman of childbearing potential not willing to use adequate contraception for the study duration
11. Patients taking anticoagulants
12. Patients who are positive serology for human immunodeficiency (HIV), hepatitis B (HBV) or hepatitis C (HCV) and syphilis
13. Patients with serious condition which can affect this study such as severe cardiovascular diseases, renal diseases, liver diseases, endocrine diseases, and cancers
14. Patients who are difficulty participating in data collection due to communication problem and serious mental illness
15. Patients are unable to come into the clinic for regular follow-up
16. Patients who had participated in other clinical trials within 3 months prior to this study.
17. Patients who the principal investigator considered inappropriate for the clinical trial due to any other reasons than those listed above.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-07-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11-07 (Actual)

PRIMARY OUTCOMES:
SPADI(Shoulder pain and disability index)Score | 24 weeks
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use.

SECONDARY OUTCOMES:
Constant-Murley score | 24 weeks
  The Constant score assesses pain, function, ROM, and strength. Pain is allotted a maximum of 15 points, activities of daily living (function)20 points, ROM 40 points, and strength 25 points. The component scores are summated to achieve a maximum possible total score of 100.
Visual Analog Scale_pain in motion | 24 weeks
Changes in the size of rotator cuff tears determined by MRI | 24 weeks
Changes in the size of rotator cuff tears determined by arthroscopy | 24 weeks
Adverse event | 24weeks

OTHER OUTCOMES:
ASES (American Shoulder and Elbow Surgeons Evaluation form) | 24 weeks
UCLA (University of California, Los Angeles) score | 24 weeks
DASH (Disabilities of the Arm, Shoulder and Hand ) | 24 weeks
WORC (Western Ontario Rotator Cuff Index) | 24 weeks
OSS (Oxford Shoulder Scores) | 24 weeks
SANE (Single Assessment Numeric Evaluation) | 24 weeks
SST (Simple Shoulder Test) | 24 weeks
Visual Analog Scale_pain at rest | 24 weeks
Visual Analog Scale_pain at night | 24 weeks
Visual Analog Scale_worst pain | 24 weeks
Visual Analog Scale_satisfaction | 24 weeks
Shoulder ROM (Forward flexion, Abduction, External rotation & Internal rotation at 0 degree) | 24 weeks
Muscle strength (lb) | 24 weeks
  The strength the supraspinatus, infraspinatus,and subscapularis was measured using a handheld electronic scale
Body weight (Kg) | 24 weeks
  To determine the overall safety of Autologous Adipose Tissue Derived Mesenchymal Stem Cells carrier using body weight
Body temperature (℃) | 24 weeks
  To determine the overall safety of Autologous Adipose Tissue Derived Mesenchymal Stem Cells carrier using body temperature
Pulse rate (beats per minute) | 24 weeks
  To determine the overall safety of Autologous Adipose Tissue Derived Mesenchymal Stem Cells carrier using pulse rate
Blood Pressure (mmHg) | 24 weeks
  To determine the overall safety of Autologous Adipose Tissue Derived Mesenchymal Stem Cells carrier using blood pressure
CBC(complete blood count) | 24 weeks
  The measures are composite.
Blood chemistry | 24 weeks
  The measures are composite.
Urinalysis | 24weeks
  The measures are composite.

CONTACTS AND LOCATIONS:
Overall Officials: Chris H. Jo, M.D., Ph.D, Principal Investigator — Joint & Spine Center, SMG-SNU Boramae Medical Center, Department of Orthopedic Surgery, Seoul National University College of Medicine
Locations (1):
- Joint & Spine Center, SMG-SNU Boramae Medical Center, Department of Orthopedic Surgery, Seoul National University College of Medicine, Seoul, South Korea